CLINICAL TRIAL: NCT05197348
Title: Spanish Adaptation of Meaning-Centered Psychotherapy for Participants With Cancer: a Protocol Study of a Randomized Control Trial
Brief Title: Spanish Meaning-Centered Psychotherapy for Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIM:2019-17
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-12

CONDITIONS: Cancer
Keywords: Meaning Centered Psychotherapy; Cancer survivors; Meaning in Life; Cognitive Behavioral Therapy; Randomized Control Trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial, efficacy Study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meaning-Centered Group Psychotherapy (MCP). (Experimental): The intervention lasts two months and includes eight sessions that follow a two-hour group format on a weekly basis. The investigators will follow the manualized MCP for patients with advanced cancer.
  Interventions: Behavioral: Meaning-Centered Group Psychotherapy (MCP).
- Cognitive Behavioral Psychotherapy (CBT). (Active Comparator): The intervention lasts two months and includes eight sessions that follow a two-hour group format on a weekly basis, with the following sessions. The investigators will follow the manualized CBT or patients with advanced cancer.
  Interventions: Behavioral: Cognitive Behavioral Psychotherapy (CBT).

INTERVENTIONS:
Behavioral: Meaning-Centered Group Psychotherapy (MCP). — The MCP program is divided into eight sessions:
  Session1: Psychoeducation about Meaning in life, Sources of Meaning, etc. Session 2: Cancer illness and meaning. Session 3: Historical Sources of Meaning (the past) Session 4: Historical Sources of Meaning (present and future). Session 5: Attitudinal Sources of Meaning. Session 6: Creative Sources of Meaning. Session 7: Experimental Sources of Meaning. Session 8: End of psychotherapy, farewell, and facing the future with hope.
  Arms: Meaning-Centered Group Psychotherapy (MCP).
Behavioral: Cognitive Behavioral Psychotherapy (CBT). — The CBT divided into eight sessions:
  Session1: Presentation of psychotherapy, establishing the goals of psychotherapy. Presentation of the participants. Updated information about psychological consequences of cancer.
  Session 2. Increase in enjoyable activities. Behavioral activation. Progressive muscle relaxation training. Slow breathing training.
  Session 3. Cognitive model of coping with cancer. Psychoeducation on negative thoughts. Training in detecting negative thoughts. Presentation of cognitive distortions Session 4. Training in cognitive restructuring techniques. Session 5. Training in problem-solving skills. Session 6. Being aware of participants needs. Self-care. Assertiveness skills training.
  Session 7. Setting goals for the future. Session 8. Summary, relapse prevention, and end of psychotherapy.
  Arms: Cognitive Behavioral Psychotherapy (CBT).

SUMMARY:
The aim of this study is to verify the efficacy of the Spanish adaptation of Meaning-Centered Psychotherapy for Spanish participants with cancer in a randomized control trial.

DETAILED DESCRIPTION:
Meaning-Centered Psychotherapy (MCP) is effective in improving meaning in life, hope, optimism, self-efficacy, well-being, and quality of life, and in reducing stress in people with cancer. However, all the studies on the application of MCP in cancer patients have been carried out in Anglo-Saxon samples. Therefore, it is necessary to adapt and verify the efficacy of MCP in populations that speak languages other than English, such as Spanish. Moreover, to expand the data supporting the efficacy of MCP for cancer patients, it would be necessary to compare MCP to other active therapies such as Cognitive Behavioral Therapy (CBT). The study has several aims: The first objective is to verify the efficacy of the MCP intervention for Spanish participants with cancer in a randomized control trial (RCT) comparing it to CBT. The second objective is to analyze the feasibility and acceptance of MCP in Spanish participants with cancer. The third objective is to analyze whether the changes produced in the Meaning in Life dimensions (presence, search, comprehension, purpose, and mattering) will predict changes in anxiety, depression, quality of life, etc.

The investigators adapted MCP for Spanish participants with cancer. The Spanish MCP is an adaptation of the MCP developed by Breitbart as an eight-session group therapy for patients with advanced cancer. This paper presents the study protocol. The study design consists of a two-arm RCT with two conditions: MCP and CBT, where participants will be randomized to one of the two groups. Participants will be adults with stage I, II, and III cancer who have completed their medical treatment (surgery, radiotherapy, or chemotherapy). Participants will be assessed at pretreatment, post-treatment, and 6-month follow-up. The intention-to-treat principle will be used when analyzing data, using mixed-effects models with full information and maximum likelihood estimation

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults with stage I, II, and III cancer who have completed their medical treatment (surgery, radiotherapy, or chemotherapy).
* Participants will have to express a need for psychological care.
* Participants will have low meaning in life.

Exclusion Criteria:

* Participants who are currently receiving another psychological or psychiatric treatment.
* Diagnosis of a serious mental disorder (schizophrenia, substance dependence, dementia, or cognitive impairment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Meaning in Life Questionnaire (MLQ) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  The MLQ is a self-reported questionnaire made up of 10 items, and it was developed to assess the two main dimensions of meaning in life: presence and search for meaning in life. The items are rated on a 7-point scale ranging from 1 (absolutely false) to 7 (absolutely true). The factors of Presence and Search were correlated (r = -.19), and internal consistency was good for Presence (.86) and Search (.87). One-month test-retest reliability coefficients were .70 for Presence and .73 for Search.
The Multidimensional Existential Meaning Scale (MEMS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  The MEMS assesses the meaning in life dimensions: Comprehension, purpose, and mattering, with a total of 15 items. Likert type responses are given on a 7-point scale (1 = Very strongly disagree; 7 = Very strongly agree). The three MEMS subscales showed adequate internal consistency: Comprehension (ϖ = 91), Purpose (ϖ = 92), and Mattering (ϖ = 86).

SECONDARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale (OASIS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  The OASIS is a five-item instrument that assesses the frequency and intensity of anxiety symptoms during the past week. In addition, it measures interference in work and academic, social, and daily life domains, as well as avoidance behaviors. The items are rated on a Likert-type scale (0-4). The psychometric properties are good in terms of internal consistency (α= 0.86), convergent and discriminant validity, and sensitivity to change (α= 0.86).
Overall Depression Severity and Impairment Scale (ODSIS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  The ODSIS is a six-item questionnaire that assesses the frequency and intensity of depression symptoms during the past week. In addition, it measures interference in work and academic, social, and daily life domains, as well as avoidance behaviors. The items are rated on a Likert-type scale (0-4). The psychometric properties are good in terms of internal consistency (α= 0.93).
Hopelessness Scale (HS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  It is a questionnaire that measures the level of hopelessness. It is made up of 20 items with dichotomous responses (True or False). It presents adequate internal consistency (α= 0.93) and has been validated in the Spanish population [39].
The Positive and Negative Affect Schedule (PANAS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  The questionnaire includes 20 adjective items, 10 assessing positive affect (PANAS-P) and 10 assessing negative affect (PANAS-N). Respondents are asked to rate the extent to which they experienced each emotion within a specified time period, using a 5-point scale (1 = Very slightly or not at all; 5 = Very much). Both affect subscales showed adequate internal consistency: PANAS-P, (α = .89) and PANAS-N (α = .91.)
Quality of life index-Spanish version (QLI) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  It is a 10-item index of perceived quality of life. It refers to physical and emotional well-being, functioning at work, personal relationships, self-independence, support in the community and from an emotional point of view, spiritual well-being, and overall perceived quality of life. The items are rated on a Likert scale (0-10) where higher scores indicate higher perceived quality of life. The psychometric properties are good for both internal consistency (α = .89) and test-retest reliability (r = 0.87).
Opinion and Expectations of Treatment Scale (OTSM) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  This scale was designed and developed by members of the research team, based on an adaptation of another opinion and expectations questionnaire. The constructs this scale assesses are: opinion, acceptance and satisfaction with the skills training program, and changes in the participants after completing each module. The questions refer to the rationale for the intervention, recommendations for the program, satisfaction with the program, and usefulness and expectations of the skills training. The items are rated on a Likert-type scale ranging from 0 "Not at all" to 10 "Very much".
Mini-Mental Adjustment to Cancer Scale. | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  This scale evaluates the different ways of coping in cancer patients. It is a self-rating questionnaire made up of 29 items that measure five dimensions of coping: fighting spirit, helplessness-hopelessness, anxious preoccupation, fatalism, and cognitive avoidance. The items are rated on a Likert scale (1-4). The Spanish version of the MINIMAC [46] showed good psychometric properties for all the subscales (fighting spirit α = .60, helplessness-hopelessness α = .82, anxious preoccupation α = .90, fatalism α = .70, and cognitive avoidance α = .80).
The Posttraumatic Growth Inventory (PTGI) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  . The PTGI is a 21-item questionnaire that assesses the perception of personal benefits in survivors of a traumatic event. A Likert response format with six categories is used, with scores ranging from 0 (no change) to 5 (very high degree of change) in a positive sense; the higher the score, the greater the change perceived. The PTGI is composed of five dimensions: Relating to others, New possibilities, Personal strength, Spiritual change and a better understanding of spiritual matters and stronger religious beliefs, and a new appreciation of life. The PTGI shows good internal consistency (α = .80).

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Llombart, Ph.D.Student, Principal Investigator — Valencian Institute of Oncology Foundation (IVO); Sandra Perez, Ph.D., Principal Investigator — University of Valencia; Veronica Guillen Botella, Ph.D., Principal Investigator — University of Valencia; Joaquin Garcia-Alandete, Ph.D., Principal Investigator — University of Valencia; Rosa Baños, Ph.D., Principal Investigator — University of Valencia; Jose Heliodoro Marco Salvador, Ph. D., Study Chair — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marco JH, Alonso S, Banos R. Meaning-making as a mediator of anxiety and depression reduction during cognitive behavioral therapy intervention in participants with adjustment disorders. Clin Psychol Psychother. 2021 Mar;28(2):325-333. doi: 10.1002/cpp.2506. Epub 2020 Sep 10. PMID 32881109
- [Background] Breitbart W, Rosenfeld B, Pessin H, Kaim M, Funesti-Esch J, Galietta M, Nelson CJ, Brescia R. Depression, hopelessness, and desire for hastened death in terminally ill patients with cancer. JAMA. 2000 Dec 13;284(22):2907-11. doi: 10.1001/jama.284.22.2907. PMID 11147988
- [Background] van der Spek N, Vos J, van Uden-Kraan CF, Breitbart W, Cuijpers P, Holtmaat K, Witte BI, Tollenaar RAEM, Verdonck-de Leeuw IM. Efficacy of meaning-centered group psychotherapy for cancer survivors: a randomized controlled trial. Psychol Med. 2017 Aug;47(11):1990-2001. doi: 10.1017/S0033291717000447. Epub 2017 Apr 4. PMID 28374663
- [Background] Vos J, Vitali D. The effects of psychological meaning-centered therapies on quality of life and psychological stress: A metaanalysis. Palliat Support Care. 2018 Oct;16(5):608-632. doi: 10.1017/S1478951517000931. Epub 2018 Sep 24. PMID 30246682
- [Background] Breitbart W, Poppito S, Rosenfeld B, Vickers AJ, Li Y, Abbey J, Olden M, Pessin H, Lichtenthal W, Sjoberg D, Cassileth BR. Pilot randomized controlled trial of individual meaning-centered psychotherapy for patients with advanced cancer. J Clin Oncol. 2012 Apr 20;30(12):1304-9. doi: 10.1200/JCO.2011.36.2517. Epub 2012 Feb 27. PMID 22370330
- [Background] Rosenfeld B, Saracino R, Tobias K, Masterson M, Pessin H, Applebaum A, Brescia R, Breitbart W. Adapting Meaning-Centered Psychotherapy for the palliative care setting: Results of a pilot study. Palliat Med. 2017 Feb;31(2):140-146. doi: 10.1177/0269216316651570. Epub 2016 Jul 21. PMID 27435603
- [Background] Lichtenthal WG, Catarozoli C, Masterson M, Slivjak E, Schofield E, Roberts KE, Neimeyer RA, Wiener L, Prigerson HG, Kissane DW, Li Y, Breitbart W. An open trial of meaning-centered grief therapy: Rationale and preliminary evaluation. Palliat Support Care. 2019 Feb;17(1):2-12. doi: 10.1017/S1478951518000925. Epub 2019 Jan 26. PMID 30683164
- [Background] Winger JG, Ramos K, Kelleher SA, Somers TJ, Steinhauser KE, Porter LS, Kamal AH, Breitbart WS, Keefe FJ. Meaning-Centered Pain Coping Skills Training: A Pilot Feasibility Trial of a Psychosocial Pain Management Intervention for Patients with Advanced Cancer. J Palliat Med. 2022 Jan;25(1):60-69. doi: 10.1089/jpm.2021.0081. Epub 2021 Aug 12. PMID 34388037
- [Derived] Marco JH, Llombart P, Romero R, Garcia-Conde A, Corral V, Guillen V, Perez S. Meaning-Centered Psychotherapy Versus Cognitive Behavioral Therapy for Cancer Survivors: A Randomized Controlled Trial☆. Behav Ther. 2024 Sep;55(5):1071-1083. doi: 10.1016/j.beth.2024.03.005. Epub 2024 Apr 10. PMID 39174266
- [Derived] Marco JH, Llombart P, Guillen V, Banos RM, Romero R, Garcia-Conde A, Perez Rodriguez S. Spanish Adaptation of Meaning-Centered Psychotherapy for Participants With Cancer: Study Protocol of a Randomized Control Trial. Front Psychiatry. 2022 Jul 7;13:892573. doi: 10.3389/fpsyt.2022.892573. eCollection 2022. PMID 35873227